CLINICAL TRIAL: NCT02793856
Title: A Phase I Clinical Trial of PD-1 Knockout Engineered T Cells Treating Patients With Advanced Non-small Cell Lung Cancer
Brief Title: PD-1 Knockout Engineered T Cells for Metastatic Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan University (Other)
Collaborators: Chengdu MedGenCell, Co., Ltd. (Industry)
Responsible Party: Principal Investigator, You Lu, Chair of Department of Thoracic Cancer, Sichuan University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MHC-001
Record Dates: First submitted 2016-05-30; First posted 2016-06-08 (Estimated); Results first posted 2020-12-21 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2020-12

CONDITIONS: Metastatic Non-small Cell Lung Cancer
Keywords: lung cancer; immune checkpoint; PD-1; CRISPR; autologous cell infusion
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A - Two cycles (Experimental): Peripheral blood lymphocytes will be collected and Programmed cell death protein 1(PDCD1) gene will be knocked out by CRISPR Cas9 in the laboratory (PD-1 Knockout T cells). The lymphocytes will be selected and expanded ex vivo and infused back into patients. Cyclophosphamide at 20mg/kg single dose will be administered 3 days i.v. before cell infusion.
  A total of 1 x 10^7/kg PD-1 Knockout T cells will be infused in one cycle. Each cycle is divided into three administrations, with 20% infused in the first administration, 30% in the second, and the remaining 50% in the third. Patients will receive a total of two cycles of treatment.
  Interventions: Drug: Cyclophosphamide; Other: PD-1 Knockout T Cells
- B- Two cycles (Experimental): Peripheral blood lymphocytes will be collected and Programmed cell death protein 1(PDCD1) gene will be knocked out by CRISPR Cas9 in the laboratory (PD-1 Knockout T cells). The lymphocytes will be selected and expanded ex vivo and infused back into patients. Cyclophosphamide at 20mg/kg single dose will be administered 3 days i.v. before cell infusion.
  A total of 2 x 10^7/kg PD-1 Knockout T cells will be infused in one cycle. Each cycle is divided into three administrations, with 20% infused in the first administration, 30% in the second, and the remaining 50% in the third. Patients will receive a total of two cycles of treatment.
  Interventions: Drug: Cyclophosphamide; Other: PD-1 Knockout T Cells
- C- Two cycles (Experimental): Peripheral blood lymphocytes will be collected and Programmed cell death protein 1(PDCD1) gene will be knocked out by CRISPR Cas9 in the laboratory (PD-1 Knockout T cells). The lymphocytes will be selected and expanded ex vivo and infused back into patients. Cyclophosphamide at 20mg/kg single dose will be administered 3 days i.v. before cell infusion.
  A total of 4 x 10^7/kg PD-1 Knockout T cells will be infused in one cycle. Each cycle is divided into three administrations, with 20% infused in the first administration, 30% in the second, and the remaining 50% in the third. Patients will receive a total of two cycles of treatment.
  Interventions: Drug: Cyclophosphamide; Other: PD-1 Knockout T Cells

INTERVENTIONS:
Drug: Cyclophosphamide — To deplete Tregs before collecting peripheral blood
  Other Names: Cytoxan
Other: PD-1 Knockout T Cells — Autologous lymphocytes are collected and PDCD1 gene is knocked out in the laboratory. Cells are selected and expanded ex vivo. Cells are infused back to the patients for treatment

SUMMARY:
This study will evaluate the safety of PD-1 knockout engineered T cells in treating metastatic non-small cell lung cancer. Blood samples will also be collected for research purposes.

DETAILED DESCRIPTION:
This is a dose-escalation study of ex-vivo knocked-out, expanded, and selected PD-1 knockout-T cells from autologous origin. Patients are assigned to 1 of 3 treatment groups to determine the maximal tolerant dose. After the lower number of cycles are considered tolerant, an arm of the next higher number of cycles will be open to next patients. Biomarkers and immunological markers are collected and analyzed as well.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically verified stage IV non-small cell lung cancer with measurable lesions (On CT: longest diameter of tumoral lesion >=10 mm, shorted diameter of lymph node >=15 mm; measurable lesions should not have been irradiated)
* Progressed after all standard treatment
* Performance score: 0-1
* Expected life span: >= 6 months
* Toxicities from prior treatment has resolved. Washout period is 4 weeks for chemotherapy, and 2 weeks for targeted therapy
* Major organs function normally
* Women at pregnant ages should be under contraception
* Willing and able to provide informed consent

Exclusion Criteria:

* Pathology is mixed type
* Emergent treatment of tumor emergency is needed
* Poor vasculature
* Coagulopathy, or ongoing thrombolytics and/or anticoagulation
* Blood-borne infectious disease, e.g. hepatitis B
* History of mandatory custody because of psychosis or other psychological disease inappropriate for treatment deemed by treating physician
* With other immune diseases, or chronic use of immunosuppressants or steroids
* Compliance cannot be expected
* Other conditions requiring exclusion deemed by physician

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-08-26 (Actual); Primary Completion 2018-08-20 (Actual); Study Completion 2020-03-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: You Lu, MD, Principal Investigator — Sichuan University
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Garon EB, Rizvi NA, Hui R, Leighl N, Balmanoukian AS, Eder JP, Patnaik A, Aggarwal C, Gubens M, Horn L, Carcereny E, Ahn MJ, Felip E, Lee JS, Hellmann MD, Hamid O, Goldman JW, Soria JC, Dolled-Filhart M, Rutledge RZ, Zhang J, Lunceford JK, Rangwala R, Lubiniecki GM, Roach C, Emancipator K, Gandhi L; KEYNOTE-001 Investigators. Pembrolizumab for the treatment of non-small-cell lung cancer. N Engl J Med. 2015 May 21;372(21):2018-28. doi: 10.1056/NEJMoa1501824. Epub 2015 Apr 19. PMID 25891174
- [Background] Brahmer J, Reckamp KL, Baas P, Crino L, Eberhardt WE, Poddubskaya E, Antonia S, Pluzanski A, Vokes EE, Holgado E, Waterhouse D, Ready N, Gainor J, Aren Frontera O, Havel L, Steins M, Garassino MC, Aerts JG, Domine M, Paz-Ares L, Reck M, Baudelet C, Harbison CT, Lestini B, Spigel DR. Nivolumab versus Docetaxel in Advanced Squamous-Cell Non-Small-Cell Lung Cancer. N Engl J Med. 2015 Jul 9;373(2):123-35. doi: 10.1056/NEJMoa1504627. Epub 2015 May 31. PMID 26028407
- [Background] Borghaei H, Paz-Ares L, Horn L, Spigel DR, Steins M, Ready NE, Chow LQ, Vokes EE, Felip E, Holgado E, Barlesi F, Kohlhaufl M, Arrieta O, Burgio MA, Fayette J, Lena H, Poddubskaya E, Gerber DE, Gettinger SN, Rudin CM, Rizvi N, Crino L, Blumenschein GR Jr, Antonia SJ, Dorange C, Harbison CT, Graf Finckenstein F, Brahmer JR. Nivolumab versus Docetaxel in Advanced Nonsquamous Non-Small-Cell Lung Cancer. N Engl J Med. 2015 Oct 22;373(17):1627-39. doi: 10.1056/NEJMoa1507643. Epub 2015 Sep 27. PMID 26412456
- [Background] Rosenberg SA, Restifo NP. Adoptive cell transfer as personalized immunotherapy for human cancer. Science. 2015 Apr 3;348(6230):62-8. doi: 10.1126/science.aaa4967. PMID 25838374
- [Background] Sharma P, Allison JP. Immune checkpoint targeting in cancer therapy: toward combination strategies with curative potential. Cell. 2015 Apr 9;161(2):205-14. doi: 10.1016/j.cell.2015.03.030. PMID 25860605
- [Background] Niu Y, Shen B, Cui Y, Chen Y, Wang J, Wang L, Kang Y, Zhao X, Si W, Li W, Xiang AP, Zhou J, Guo X, Bi Y, Si C, Hu B, Dong G, Wang H, Zhou Z, Li T, Tan T, Pu X, Wang F, Ji S, Zhou Q, Huang X, Ji W, Sha J. Generation of gene-modified cynomolgus monkey via Cas9/RNA-mediated gene targeting in one-cell embryos. Cell. 2014 Feb 13;156(4):836-43. doi: 10.1016/j.cell.2014.01.027. Epub 2014 Jan 30. PMID 24486104
- [Derived] Lu Y, Xue J, Deng T, Zhou X, Yu K, Deng L, Huang M, Yi X, Liang M, Wang Y, Shen H, Tong R, Wang W, Li L, Song J, Li J, Su X, Ding Z, Gong Y, Zhu J, Wang Y, Zou B, Zhang Y, Li Y, Zhou L, Liu Y, Yu M, Wang Y, Zhang X, Yin L, Xia X, Zeng Y, Zhou Q, Ying B, Chen C, Wei Y, Li W, Mok T. Safety and feasibility of CRISPR-edited T cells in patients with refractory non-small-cell lung cancer. Nat Med. 2020 May;26(5):732-740. doi: 10.1038/s41591-020-0840-5. Epub 2020 Apr 27. PMID 32341578
- [Derived] Yi L, Li J. CRISPR-Cas9 therapeutics in cancer: promising strategies and present challenges. Biochim Biophys Acta. 2016 Dec;1866(2):197-207. doi: 10.1016/j.bbcan.2016.09.002. Epub 2016 Sep 15. PMID 27641687

RESULTS

PARTICIPANT FLOW:
Groups:
- Pre-A-One Cycle: Peripheral blood lymphocytes will be collected and Programmed cell death protein 1(PDCD1) gene will be knocked out by CRISPR Cas9 in the laboratory (PD-1 Knockout T cells). The lymphocytes will be selected and expanded ex vivo and infused back into patients. Cyclophosphamide at 20mg/kg single dose will be administered 3 days i.v. before cell infusion.
  A total of 2 x 10^7/kg PD-1 Knockout T cells will be infused in one cycle which is divided into three administrations, with 20% infused in the first administration, 30% in the second, and the remaining 50% in the third. Patients will receive a total of one cycle of treatment.
  Cyclophosphamide: To deplete Tregs before collecting peripheral blood
  PD-1 Knockout T Cells: Autologous lymphocytes are collected and PDCD1 gene is knocked out in the laboratory. Cells are selected and expanded ex vivo. Cells are infused back to the patients for treatment
- A - Two Cycles: Peripheral blood lymphocytes will be collected and Programmed cell death protein 1(PDCD1) gene will be knocked out by CRISPR Cas9 in the laboratory (PD-1 Knockout T cells). The lymphocytes will be selected and expanded ex vivo and infused back into patients. Cyclophosphamide at 20mg/kg single dose will be administered 3 days i.v. before cell infusion.
  A total of 1 x 10^7/kg PD-1 Knockout T cells will be infused in one cycle. Each cycle is divided into three administrations, with 20% infused in the first administration, 30% in the second, and the remaining 50% in the third. Patients will receive a total of two cycles of treatment.
  Cyclophosphamide: To deplete Tregs before collecting peripheral blood
  PD-1 Knockout T Cells: Autologous lymphocytes are collected and PDCD1 gene is knocked out in the laboratory. Cells are selected and expanded ex vivo. Cells are infused back to the patients for treatment
- B- Two Cycles: Peripheral blood lymphocytes will be collected and Programmed cell death protein 1(PDCD1) gene will be knocked out by CRISPR Cas9 in the laboratory (PD-1 Knockout T cells). The lymphocytes will be selected and expanded ex vivo and infused back into patients. Cyclophosphamide at 20mg/kg single dose will be administered 3 days i.v. before cell infusion.
  A total of 2 x 10^7/kg PD-1 Knockout T cells will be infused in one cycle. Each cycle is divided into three administrations, with 20% infused in the first administration, 30% in the second, and the remaining 50% in the third. Patients will receive a total of two cycles of treatment.
  Cyclophosphamide: To deplete Tregs before collecting peripheral blood
  PD-1 Knockout T Cells: Autologous lymphocytes are collected and PDCD1 gene is knocked out in the laboratory. Cells are selected and expanded ex vivo. Cells are infused back to the patients for treatment
- C- Two Cycles: Peripheral blood lymphocytes will be collected and Programmed cell death protein 1(PDCD1) gene will be knocked out by CRISPR Cas9 in the laboratory (PD-1 Knockout T cells). The lymphocytes will be selected and expanded ex vivo and infused back into patients. Cyclophosphamide at 20mg/kg single dose will be administered 3 days i.v. before cell infusion.
  A total of 4 x 10^7/kg PD-1 Knockout T cells will be infused in one cycle. Each cycle is divided into three administrations, with 20% infused in the first administration, 30% in the second, and the remaining 50% in the third. Patients will receive a total of two cycles of treatment.
  Cyclophosphamide: To deplete Tregs before collecting peripheral blood
  PD-1 Knockout T Cells: Autologous lymphocytes are collected and PDCD1 gene is knocked out in the laboratory. Cells are selected and expanded ex vivo. Cells are infused back to the patients for treatment
Period: Overall Study
Arm/Group | Pre-A-One Cycle | A - Two Cycles | B- Two Cycles | C- Two Cycles
Started | 2 | 4 | 3 | 3
Completed | 2 | 4 | 3 | 3
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Pre-A-One Cycle: Peripheral blood lymphocytes will be collected and Programmed cell death protein 1(PDCD1) gene will be knocked out by CRISPR Cas9 in the laboratory (PD-1 Knockout T cells). The lymphocytes will be selected and expanded ex vivo and infused back into patients. Cyclophosphamide at 20mg/kg single dose will be administered 3 days i.v. before cell infusion.
  A total of 2 x 10^7/kg PD-1 Knockout T cells will be infused in one cycle. Each cycle is divided into three administrations, with 20% infused in the first administration, 30% in the second, and the remaining 50% in the third. Patients will receive a total of one cycle of treatment.
  Cyclophosphamide: To deplete Tregs before collecting peripheral blood
  PD-1 Knockout T Cells: Autologous lymphocytes are collected and PDCD1 gene is knocked out in the laboratory. Cells are selected and expanded ex vivo. Cells are infused back to the patients for treatment
- Total: Total of all reporting groups
Arm/Group | Pre-A-One Cycle | A - Two Cycles | B- Two Cycles | C- Two Cycles | Total
Number analyzed (Participants) | 2 | 4 | 3 | 3 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 2 | 3 | 10
  >=65 years | 0 | 1 | 1 | 0 | 2
Age, Continuous [Median (Full Range); unit: years] | 55.5 [48 to 63] | 56 [48 to 66] | 55 [31 to 68] | 53 [47 to 61] | 54.5 [31 to 68]
Age, Continuous [Mean (Full Range); unit: years] | 55.5 [48 to 63] | 56 [48 to 66] | 55 [31 to 68] | 53 [47 to 61] | 54.5 [31 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2 | 0 | 4
  Male | 2 | 2 | 1 | 3 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 4 | 3 | 3 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 2 | 4 | 3 | 3 | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events and/or Dose Limiting Toxicities as a Measure of Safety and Tolerability of Dose of PD-1 Knockout T Cells Using Common Terminology Criteria for Adverse Events (CTCAE v4.0) in Patients
Time Frame: Dose Escalation - Approximately 6 months
Measure: Count of Participants; unit: Participants
Groups:
- Pre-A Cohort; A Cohort; B Cohort; C Cohort: All adverse events are grade 1-2.
Arm/Group | Pre-A Cohort | A Cohort | B Cohort | C Cohort
Number analyzed (Participants) | 2 | 4 | 3 | 3
Participants | 2 | 4 | 3 | 2

2. Secondary Outcome: Number of Patients With Overall Response
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR."
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Groups:
- Pre-A Cohort: In Pre-A Cohort, all patient were assessed per RECIST v1.1
- A Cohort: In A Cohort, 3 patients were assessed per RECIST v1.1. One patient was unavailable for tumor response assessment due to early withdrawal.
- B Cohort: In B Cohort, all patients were assessed per RECIST v1.1.
- C Cohort: In C Cohort, all patients were assessed per RECIST v1.1.
Arm/Group | Pre-A Cohort | A Cohort | B Cohort | C Cohort
Number analyzed (Participants) | 2 | 3 | 3 | 3
Participants | 0 | 0 | 0 | 0

3. Secondary Outcome: Number of Patients With Disease Control at 8 Weeks
Description: Response will be evaluated according to RECIST v1.1 for target lesions at Week 8：Complete Response (CR), Disappearance of all extranodal target lesions; Partial Response (PR) ≥ 30% decrease in the sum of diameters of target lesions; Stable Disease (SD) Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD; Disease control = CR +PR+SD
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Pre-A Cohort: In Pre-A Cohort, all two patients were assessed per RECIST v1.1.
- A Cohort: 3 patients were assessed per RECIST v1.1. One patient was unavailable for tumor response assessment due to early withdrawal.
- C Cohort: All patients were assessed per RECIST v1.1.
Arm/Group | Pre-A Cohort | A Cohort | B Cohort | C Cohort
Number analyzed (Participants) | 2 | 3 | 3 | 3
Participants | 1 | 0 | 1 | 0

4. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: The time from the date of first edited T cell infusion to the date of disease progression or death due to any reason.
Measure: Median (95% Confidence Interval); unit: weeks
Groups:
- A Cohort; C Cohort: All patients were assessed per RECIST v1.1.
Arm/Group | Pre-A Cohort | A Cohort | B Cohort | C Cohort
Number analyzed (Participants) | 2 | 4 | 3 | 3
weeks | 11.7 [5.6 to 17.7] | 8.0 [7.3 to 8.4] | 8.1 [7.4 to 75.7] | 6.1 [5.0 to 8.1]

5. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time interval from date of first edited T cell infusion to the date of death due to any reason
Time Frame: The duration from date of first edited T cell infusion to the date of death due to any reason
Measure: Median (95% Confidence Interval); unit: weeks
Groups:
- Pre-A Cohort: In Pre-A Cohort, two patients were followed up.
- A Cohort; C Cohort: All patients were followed up.
- B Cohort: In B Cohort, all patients were followed up.
Arm/Group | Pre-A Cohort | A Cohort | B Cohort | C Cohort
Number analyzed (Participants) | 2 | 4 | 3 | 3
weeks | 47.5 [42.6 to 52.4] | 51.4 [13.4 to 116] | 32.6 [24.4 to 97.7] | 51.6 [21 to 96.7]

6. Secondary Outcome: Number of Participants With Genes Mutations in Peripheral Blood Circulating Tumor DNA (ctDNA)
Description: Driver genes mutaion stauts of Participants in ctDNA from peripheral blood were assessed by next generation sequencing (NGS), to explore the positive rate of sepicif driver genes (e.g. EGFR, ALK, ROS1, etc.) and the relationship between gene mutation status and clinical response
Time Frame: Baseline
Population: Only three patients were detected with EGFR mutations. Correlation between driver gene mutations with clinical outcome were not analyzed due to limited data. EGFR positive rate was showed in outcome measure data table.
Measure: Count of Participants; unit: Participants
Groups:
- Pre-A Cohort; A Cohort; B Cohort; C Cohort: All patients were tested for gene mutation status in ctDNA at baseline
Arm/Group | Pre-A Cohort | A Cohort | B Cohort | C Cohort
Number analyzed (Participants) | 2 | 4 | 3 | 3
Participants | 0 | 1 | 1 | 1

7. Secondary Outcome: Interleukin-6 Change in the Peripheral Blood.
Description: Peripheral Interleukin-6 level at different timepoint (Baseline, 1 month and 3 month) was measured using rate nephelometry
Time Frame: Baseline, 1 month and 3 month
Population: One patients did not provide blood sample due to early withdrawal; blood samples of 8 patients were only collected at baseline and month 1 due to PD before month 3
Measure: Median (95% Confidence Interval); unit: pg/ml
Groups:
- Pre-A Cohort: In Pre-A Cohort, one patient provided blood smaple at baseline, month 1 and month 3, the other patient provided blood sample only at baseline and month 1.
- A Cohort: Three patients were collected blood at baseline and month 1. The other patient's sample was not collected owing to early withdrawal from the trial. All patients had relapsed disease before month 3 and were not able to samples at month 3.
- B Cohort: In B Cohort, One patient's blood was collected at baseline, month 1 and month 3. The other two patients' sample were collected only at baseline and month 1 owing to PD before month 3.
- C Cohort: In C Cohort, One patient's blood was collected blood at baseline, month 1 and month 3. The other two patients' blood were only collected blood at baseline and month 1, owing to PD before month 3.
Arm/Group | Pre-A Cohort | A Cohort | B Cohort | C Cohort
Number analyzed (Participants) | 2 | 3 | 3 | 3
pg/ml
  baseline | 10.68 [8.98 to 12.38] | 3.27 [2.62 to 61.87] | 51.97 [8.09 to 67.09] | 10.59 [10.28 to 11.45]
  1 month | 12.9 [1.5 to 24.3] | 4.37 [2.39 to 90.17] | 23.92 [5.58 to 137.1] | 14.77 [8.48 to 26.17]
  3 month: number analyzed (Participants) | 1 | 0 | 1 | 1
  3 month | 18.45 [18.45 to 18.45] |  | 4.03 [4.03 to 4.03] | 12.49 [12.49 to 12.49]

8. Secondary Outcome: Interleukin-10 Change in the Peripheral Blood.
Description: Peripheral Interleukin-10 level at different timepoint (Baseline, 1 month and 3 month) was measured using chemiluminescence.
Time Frame: Baseline, 1 month and 3 month
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: pg/ml
Groups:
- Pre-A Cohort: In Pre-A Cohort, one patient's blood was collected blood at baseline, month 1 and month 3, the other patient's blood was collected at baseline and month 1.
- A Cohort: Three patients' samples were collected at baseline and month 1. The other patient's sample was not collected owing to early withdrawal from the trial. All patients had relapsed disease before month 3 and did not provide samples at month 3
- B Cohort: In B Cohort, One patient's sample was collected at baseline, month 1 and month 3. The other two patients' samples were collected only at baseline and month 1, owing to PD before month 3.
- C Cohort: In C Cohort, one patient's sample was collected at baseline, month 1 and month 3. The other two patients' samples were collected only at baseline and month 1, owing to PD before month 3.
Arm/Group | Pre-A Cohort | A Cohort | B Cohort | C Cohort
Number analyzed (Participants) | 2 | 3 | 3 | 3
pg/ml
  baseline | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00]
  1 month | 5.00 [5.00 to 5.00] | 5.00 [5.00 to 5.00] | 19.05 [7.3 to 30.8] | 5.00 [5.00 to 5.00]
  3 month: number analyzed (Participants) | 1 | 0 | 1 | 1
  3 month | 5.00 [5.00 to 5.00] |  | 27.10 [27.10 to 27.10] | 5.00 [5.00 to 5.00]

9. Secondary Outcome: Tumor Necrosis Factor-a Change in the Peripheral Blood.
Description: Peripheral Tumor Necrosis Factor-a level at different timepoint (Baseline, 1 month and 3 month) was measured using chemiluminescence.
Time Frame: Baseline, 1 month and 3 month
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: pg/ml
Groups:
- Pre-A Cohort: In Pre-A Cohort, one patient's blood was collected at baseline, month 1 and month 3, the other patient's blood was collected only at baseline and month 1.
- A Cohort: Three patients provided blood samples at baseline and month 1. The other patient's sample was not collected owing to early withdrawal from the trial. All patients had relapsed disease before month 3 and were not able to provide samples at month 3
- B Cohort: In B Cohort, one patient's sample was collected at baseline, month 1 and month 3. The other two patients' sample were collected only at baseline, month 1 owing to PD before month 3.
- C Cohort: In C Cohort, one patient's sample was collected at baseline, month 1 and month 3. The other two patients' sample were collected only at baseline, month 1 owing to PD before month 3.
Arm/Group | Pre-A Cohort | A Cohort | B Cohort | C Cohort
Number analyzed (Participants) | 2 | 3 | 3 | 3
pg/ml
  baseline | 13.84 [7.97 to 19.7] | 6.07 [5.61 to 8.53] | 8.89 [5.30 to 8.92] | 5.06 [4.01 to 6.28]
  1 month | 10.68 [7.65 to 13.7] | 7.84 [5.74 to 7.92] | 10.40 [4.2 to 11.9] | 16.4 [6.31 to 27.70]
  3 month: number analyzed (Participants) | 1 | 0 | 1 | 1
  3 month | 6.97 [6.97 to 6.97] |  | 10.90 [10.90 to 10.90] | 11.70 [11.70 to 11.70]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 2 years.
Description: Grade 1/2 treatment-related adverse events (AEs) occurred in 11 of the 12 patients and There were no grade ≥3 treatment-related AEs
Groups:
- Pre-A Cohort; C Cohort: Grade 1/2 treatment-related adverse events (AEs) occurred in 2 patients.
- A Cohort: Grade 1/2 treatment-related adverse events (AEs) occurred in 4 patients.
- B Cohort: Grade 1/2 treatment-related adverse events (AEs) occurred in 3 patients.
Arm/Group | Pre-A Cohort | A Cohort | B Cohort | C Cohort
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/4 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/4 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 2/2 | 4/4 | 3/3 | 2/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pre-A Cohort (N=2) | A Cohort (N=4) | B Cohort (N=3) | C Cohort (N=3)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Arthralgia (Immune system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Premature beats (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Increased AST (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 | 2 (2) | 0
Hypertension (General disorders) | 1 (1) | 0 | 0 | 0
Increased ALT (Immune system disorders) | 1 (1) | 0 | 0 | 0
Fever (General disorders) | 0 | 0 | 2 (2) | 0
Hyperhidrosis (General disorders) | 0 | 0 | 1 (1) | 0
Infusion-related reaction (General disorders) | 0 | 1 (1) | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 (1) | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 (1) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-04): https://cdn.clinicaltrials.gov/large-docs/56/NCT02793856/Prot_SAP_000.pdf